CLINICAL TRIAL: NCT01012349
Title: Efficacy and Safety Clinical Trial of the Combination of Acetylsalicylic Acid, Sodium Bicarbonate and Citric Acid, Produced by Geolab Pharmaceutical Industries Ltd., Compared to Acetylsalicylic Acid (Aspirin ® - Bayer) in Patients With Episodic Tension-type Headache.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AASGEO0809; Version 2
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2010-10

CONDITIONS: Treatment of Episodic Tension Headache
MeSH Terms: interventions — Sodium Bicarbonate; Citric Acid; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): Administration of GeoLab Association (acetylsalicylic acid, sodium bicarbonate and citric acid)
  Interventions: Drug: Association: acetylsalicylic acid (500mg), sodium bicarbonate (1625) and citric acid (965)
- Comparator (Active Comparator): Acetylsalicylic acid - (Aspirin - Bayer)
  Interventions: Drug: Aspirin - Bayer

INTERVENTIONS:
Drug: Association: acetylsalicylic acid (500mg), sodium bicarbonate (1625) and citric acid (965) — 1 tablet in an episody of headache
  Arms: Test
Drug: Aspirin - Bayer — 1 tablet in an episody of headache (Aspirin 500mg)
  Arms: Comparator

SUMMARY:
This study aims is to evaluate, two hours after a single administration, the rate of sustained response produced by the association Geolab consisting of acetylsalicylic acid, sodium bicarbonate and anhydrous citric acid - oral powder, with the active comparator acetylsalicylic acid (Aspirin ® -- Bayer) - a simple tablet for the treatment of acute pain in patients with mild to moderate CTTE, using for both the visual analog scale pain - VAS.

DETAILED DESCRIPTION:
The secondary objectives of the study are to evaluate:

* Modification of gastric pH after administration of drugs by measuring with gastroesophageal pH Monitor, comparing the results between the groups;
* The incidence of administration of rescue medications, through the accounts of patients and researchers, comparing the results between the groups;
* The percentage of improvement in time 30, 60, 90 and 120 minutes after administration, using the visual analog scale (VAS), comparing the results between the groups;
* Evaluate the gastric symptoms before and after treatment by clinical investigation of patients, comparing the results between the groups;
* Evaluate the change in associated symptoms (photophobia, phonophobia, nausea, vomiting), using 4-point scale (0 - absent 1 - mild 2 - moderate 3 - severe), comparing the results between the groups;
* Assess the quantitative and qualitative parameters related to adverse reactions, comparing the results between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Agreed to participate in the study expressed by signing the two copies of the informed consent and informed consent (IC) after approved by the IRB;
* Minimum age of 18 years;
* Clinical history of TTH, according to the criteria of the International Classification of Headache of the International Headache Society, in face of crisis.

Exclusion Criteria:

* Headache, migraine
* Chronic Tension-Type Headache (CTTH)
* Altered mental status
* Vital signs changed
* established or suspected pregnancy and lactation
* History of allergy to components of study drugs
* Current treatment with methotrexate
* Current treatment with Antinauseants
* Current treatment with anticoagulants such as heparin or coumarin-derivative
* gastric or duodenal disorders, chronic or recurrent active
* Liver and kidney disease severe
* Use of medications that have drug interactions with AAS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-05 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the rate of sustained response (percentage of subjects who have no pain) two hours after the drug administration. | 0, 30, 60, 90 and 120 minutes

SECONDARY OUTCOMES:
• Reduction of associated symptoms (photophobia, phonophobia, nausea, vomiting); • Symptoms stomach before and after treatment • Change in gastric pH after administration; • Incidence of administration of rescue medications; • Change in pain | 30, 60, 90 and 120 minutes after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Lal Clinica Pesquisa E Desenvolvimento Ltda, Valinhos, São Paulo, Brazil